CLINICAL TRIAL: NCT04703686
Title: A Phase II Trial Evaluating Glofitamab, a Bispecific CD3xCD20 Antibody for Relapse/Refractory Lymphomas After CAR T-cells Therapy
Brief Title: Treatment by a Bispecific CD3xCD20 Antibody for Relapse/Refractory Lymphomas After CAR T-cells Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BiCAR
Record Dates: First submitted 2021-01-04; First posted 2021-01-11 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Diffuse Large B-Cell Lymphoma Refractory; Refractory Indolent Adult Non-Hodgkin Lymphoma; Refractory Transformed B-cell Non-Hodgkin Lymphoma; Refractory Primary Mediastinal Large B-Cell Cell Lymphoma; Refractory Mantle Cell Lymphoma
Keywords: Post Car T-cells therapy
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — obinutuzumab; glofitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obinutuzumab + RO7082859 (Experimental)
  Interventions: Drug: Obinutuzumab; Drug: RO7082859

INTERVENTIONS:
Drug: Obinutuzumab — 1000mg - prephase - one infusion at D-3
  Other Names: gazyva
Drug: RO7082859 — 2.5 mg D1C1, 10 mg D3C1, then 30 mg D8C1 and D1 every 21 days (C2-C11, D1C2 starts 14 days after D1C1)
  Other Names: glofitamab

SUMMARY:
This study is a multicenter phase II trial including 2 cohorts of patients in Refractory/Relapse disease at least 1 month after CAR T-cells therapy:

* cohort 1: DLBCL patients
* cohort 2: PMBL, mantle cell lymphoma, transformed indolent NHL (t-iNHL) or iNHL CAR T-cells Refractory/Relapse status will be determined by PET-CT central review allowing inclusion in this trial.

Patients enrolled will then receive a pre-phase of obinutuzumab followed by experimental treatment:11 cycle of glofitamab.

The primary objective of the study is to assess the anti-lymphoma activity of glofitamab, a bispecific CD3xCD20 monoclonal antibody in patients with relapse/refractory DLBCL (cohort 1) disease after anti-CD19 CAR T-cells therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received CAR T-cells therapy for R/R DLBCL (cohort 1) or R/R PMBL, mantle cell lymphoma, t-iNHL or iNHL (cohort 2), at least 1 month ago
2. Patients who are not, at least in partial metabolic response from 1 month after CAR T-cells infusion (i.e no metabolic response or first metabolic progressive disease or first relapse from 1 month after CAR T-cells infusion)
3. First metabolic progression, first relapse or no metabolic response after CAR T-cells infusion must be confirmed by PET-CT central review for enrollment
4. DLBCL with demonstrated lymphoma cells-expressing CD20 at relapse post CAR T-cells as demonstrated by biopsy before enrollment (cohort 1 only)
5. Aged 18 years or more with no upper age limit
6. ECOG performance status 0 or 1
7. Bi-dimensionally measurable disease defined by at least one single node or tumor lesion > 1.5 cm assessed by CT scan, or PET-CT with at least one hypermetabolic lesion
8. No persistant CAR-T neurotoxicity symptoms or previous experience during CAR T-cells therapy of neurotoxicity grade > 3
9. Adverse events from prior anti-cancer therapy must have resolved to Grade ≤ 1 (hematological toxicities excepted)
10. Adequate liver function: Total bilirubin ≤ 1.5 x ULN; Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x ULN Note: Patients with documented history of Gilbert's Syndrome and in whom total bilirubin elevations are accompanied by elevated indirect bilirubin are eligible)
11. Adequate hematological function: Neutrophil count of ≥ 1.0 G/L; Platelet count of ≥ 50 G/L (and platelet transfusion free within 14 days prior to administration of obinutuzumab); Hemoglobin (Hb) ≥ 8.0 g/dL (transfusion free within 21 days prior to administration of obinutuzumab) Note: patients who do not meet the above hematologic criteria, due to extensive tumor involvement in the marrow may be enrolled into the trial after the demonstration of involvement and consultation with the LYSARC. Please consult the LYSARC on the need for transfusion support within 21 days of obinutuzumab
12. Adequate renal function: creatinine clearance (CrCl) calculated by MDRD/cockcroft -Gault formula of ≥ 30 mL/min
13. Negative serum or urinary pregnancy test within 7 days prior to study treatment in women of childbearing potential
14. Negative serologic or PCR test results for acute or chronic HBV infection Note: Patients whose HBV infection status cannot be determined by serologic test results must be negative for HBV by PCR to be eligible for study participation
15. Negative test results for HCV and HIV Note: Patients who are positive for HCV antibody must be negative for HCV by PCR to be eligible for study participation
16. Patients must agree to either remain completely abstinent or to use two effective contraceptive methods* until:

    * If the patient is a male: at least 3 months after pre-treatment with obinutuzumab or 2 months after the last dose of glofitamab, whichever is longer, Men must refrain from donating sperm during this same period
    * If patient is a female of childbearing potential: until at least 18 months after pre-treatment with obinutuzumab or 2 months after the last dose of glofitamab, whichever is longer
17. Patient must be willing and able to comply with protocol-mandated hospitalization upon administration of the first dose of glofitamab. Patient must also be willing to comply with all study-related procedures.
18. Signed written informed consent
19. Life expectancy ≥ 3 months
20. Patient covered by any social security system
21. Patient who understands and speaks one of the country official languages

Exclusion Criteria:

1. Previously known CD20 negative status, excepted if a new biopsy for cohort 1 or biopsy or cytometry analysis for cohort 2 proving a CD20 positive status is available before enrollment
2. Patients with CLL, Richter and Burkitt lymphoma
3. Patients relapsing or progressing within 1 months (30 days) after CAR T-cells therapy
4. History of treatment-emergent immune-related adverse events associated with prior immunotherapeutic agents, as follows:

   * Grade ≥ 3 adverse events with the exception of Grade 3 endocrinopathy managed with replacement therapy
   * Grade 1-2 adverse events that did not resolve to baseline after treatment discontinuation
5. Current or past history of detectable cerebrospinal fluid lymphoma cells, or with a history of CNS lymphoma localization or primary CNS lymphoma
6. Current or past history of cerebral disorders
7. Any serious psychiatric illness that would prevent the subject from signing the informed consent form.
8. Patients with history of macrophage activation syndrome (MAS) / hemophagocytic lymphohistiocytosis (HLH)
9. Patients with known acute infection or reactivation of a latent infection, whether bacterial, viral (including, but not limited to, EBV, cytomegalovirus (CMV), hepatitis B, hepatitis C, and HIV), fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics this pertains to completion of last course of antibiotic treatment) in 2 week prior to enrollment
10. LVEF < 40% as determined by echocardiography or multiple uptake gated acquisition (MUGA) scan or significant cardiovascular disease such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina)
11. Any serious active disease or co-morbid medical condition
12. Clinically significant history of liver disease or cirrhosis
13. Prior history of malignancies other than lymphoma unless the subject has been free of the disease for ≥ 3 years. Exceptions will be allowed for patients with non-melanoma skin tumors (basal cell or squamous cell carcinoma of the skin) or any surgically removed stage 0 (in situ) carcinoma
14. Prior solid organ transplantation
15. Prior allogeneic SCT
16. Autologous SCT within 100 days prior to obinutuzumab infusion
17. Current uncontrolled autoimmune disease Note: History of autoimmune disease currently controlled and stable is acceptable for such therapy. See detailed description below*
18. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
19. Major surgery or significant traumatic injury < 28 days prior to the obinutuzumab infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
20. Administration of a live, attenuated vaccine within 4 weeks before obinutuzumab infusion
21. Treatment between infusion of CAR T-cells and pre-phase (i.e. obinutuzumab infusion on C1/D-3): with standard radiotherapy, systemic immunotherapeutic agents, any chemotherapeutic agent, any systemic immunosuppressive medications or treatment with any other investigational anti-cancer agent (defined as treatment for which there is currently no regulatory authority approved indication) Note: with the exception of corticosteroid treatment < 25 mg/day prednisone or equivalent. Inhaled and topical steroids are permitted
22. Patient with history of confirmed progressive multifocal leukoencephalopathy (PML)
23. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
24. History of illicit drug or alcohol abuse within 12 months prior to enrollment
25. Person deprived of his/her liberty by a judicial or administrative decision
26. Inability to comply with protocol mandated hospitalization and restrictions
27. Adult person under legal protection
28. Adult person unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness
29. Pregnant or breast-feeding or intending to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 4 years
  Overall survival will be measured from the date of C1D1 of glofitamab to the date of death from any cause. Alive patients will be censored at the date of last contact

SECONDARY OUTCOMES:
Metabolic response rates according to Lugano classification | At the end of Cycle 2 (1st cycle of 14 days and subsequent cycles of 21 days)
  Response will be assessed by local and central review by PET scan according to Lugano classification
Metabolic response rates according to Lugano classification | At the end of Cycle 6 (1st cycle of 14 days and subsequent cycles of 21 days)
  Response will be assessed by local and central review by PET scan according to Lugano classification
Metabolic response rates according to Lugano classification | At the end of Cycle 9 (1st cycle of 14 days and subsequent cycles of 21 days)
  Response will be assessed by local and central review by PET scan according to Lugano classification
Metabolic response rates according to Lugano classification | At the end of Cycle 11 (1st cycle of 14 days and subsequent cycles of 21 days)
  Response will be assessed by local and central review by PET scan according to Lugano classification
Progression Free Survival (PFS) | At the end of Cycle 2 (1st cycle of 14 days and subsequent cycles of 21 days)
  PFS is defined as the time from enrollment into the study to the first observation of documented disease progression based on central review or death due to any cause
Progression Free Survival (PFS) | At the end of Cycle 4 (1st cycle of 14 days and subsequent cycles of 21 days)
  PFS is defined as the time from enrollment into the study to the first observation of documented disease progression based on central review or death due to any cause
Progression Free Survival (PFS) | At the end of Cycle 6 (1st cycle of 14 days and subsequent cycles of 21 days)
  PFS is defined as the time from enrollment into the study to the first observation of documented disease progression based on central review or death due to any cause
Progression Free Survival (PFS) | At the end of Cycle 9 (1st cycle of 14 days and subsequent cycles of 21 days)
  PFS is defined as the time from enrollment into the study to the first observation of documented disease progression based on central review or death due to any cause
Progression Free Survival (PFS) | At the end of Cycle 11 (1st cycle of 14 days and subsequent cycles of 21 days)
  PFS is defined as the time from enrollment into the study to the first observation of documented disease progression based on central review or death due to any cause
Duration of Response (DoR) | At the end of Cycle 2 (1st cycle of 14 days and subsequent cycles of 21 days)
  DoR is defined from the time of first CMR or PMR (according to Lugano criteria) to the date of first documented disease progression, relapse or death from any cause. If a subject has not progressed or died, DoR will be censored at the date of tumor assessment
Duration of Response (DoR) | At the end of Cycle 4 (1st cycle of 14 days and subsequent cycles of 21 days)
  DoR is defined from the time of first CMR or PMR (according to Lugano criteria) to the date of first documented disease progression, relapse or death from any cause. If a subject has not progressed or died, DoR will be censored at the date of tumor assessment
Duration of Response (DoR) | At the end of Cycle 6 (1st cycle of 14 days and subsequent cycles of 21 days)
  DoR is defined from the time of first CMR or PMR (according to Lugano criteria) to the date of first documented disease progression, relapse or death from any cause. If a subject has not progressed or died, DoR will be censored at the date of tumor assessment
Duration of Response (DoR) | At the end of Cycle 9 (1st cycle of 14 days and subsequent cycles of 21 days)
  DoR is defined from the time of first CMR or PMR (according to Lugano criteria) to the date of first documented disease progression, relapse or death from any cause. If a subject has not progressed or died, DoR will be censored at the date of tumor assessment
Duration of Response (DoR) | At the end of Cycle 11 (1st cycle of 14 days and subsequent cycles of 21 days)
  DoR is defined from the time of first CMR or PMR (according to Lugano criteria) to the date of first documented disease progression, relapse or death from any cause. If a subject has not progressed or died, DoR will be censored at the date of tumor assessment
Quality of Life - QLQ-C30 | at day 1
  Quality of Life scale measurements will be the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30),
Quality of Life - FACT-Lym LymS | at day 1
  Quality of Life scale measurements will be the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym LymS) subscale
Quality of Life - QLQ-C30 | At Cycle 2 Day 1 (1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Quality of Life - FACT-Lym LymS | At Cycle 2 Day 1 (1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym LymS) subscale
Quality of Life - EORTC QLQ-C30 | At Cycle 3 Day 1(1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Quality of Life _ FACT-Lym LymS | At Cycle 3 Day 1(1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym LymS) subscale
Quality of Life - QLQ-C30 | At cycle 5 day 1 (1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Quality of Life _ FACT-Lym LymS | At cycle 5 day 1 (1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym LymS) subscale
Quality of Life _ QLQ-C30 | At Cycle 7 Day 1(1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Quality of Life _ FACT-Lym LymS | At Cycle 7 Day 1 (1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym LymS) subscale
Quality of Life _ QLQ-C30 | At Cycle 9 Day 1(1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Quality of Life _ FACT-Lym LymS | At Cycle 9 Day 1(1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym LymS) subscale
Quality of Life _ QLQ-C30 | At Cycle 11 Day 1(1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Lifescale measurements will be the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Quality of Life _ FACT-Lym LymS | At Cycle 11 Day 1(1st cycle of 14 days and subsequent cycles of 21 days)
  Quality of Life scale measurements will be the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym LymS) subscale
number of Serious Adverse Events | from the date of first informed consent signature to 30 days after last administration of study drugs
Best metabolic response assessed by local review | after 11 cycles (1st cycle of 14 days and subsequent cycles of 21 days)
Best metabolic response assessed by central review | after 11 cycles (1st cycle of 14 days and subsequent cycles of 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Cartron, MD,PhD, Study Chair — Lymphoma Study Association; Pierre Sesques, MD, Study Chair — Lymphoma Study Association
Locations (15):
- France (15):
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - CHRU Lille - Hôpital Claude Huriez, Lille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hôpital Saint Louis, Paris
  - APHP - Hôpital de la Pitiè Salpetrière, Paris
  - APHP - Hôpital Saint Antoine, Paris
  - CHU de Bordeaux - Hôpital Haut Leveque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - IUCT Oncopole, Toulouse
  - CHU de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No